CLINICAL TRIAL: NCT06100588
Title: The Classification of Myofascial Headache: a Cross-sectional Study. the Added Value of Dry Needling in the Treatment of Myofascial Headache: a Randomized Controlled Trial.
Brief Title: The Classification and Treatment of Myofascial Headache: a Cross-sectional Study and Randomized Controlled Trial.
Acronym: COMPHAS_RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2023-0377
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Tension-Type Headache; Cervicogenic Headache; Myofascial Headache
Keywords: Dry Needling; Manual Therapy; Headache
MeSH Terms: conditions — Tension-Type Headache; Post-Traumatic Headache; Headache | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Particpants will be randomly assigned to either of the following groups:
  * Treatment with manual therapy;
  * Treatment with manual therapy in combination with dry needling.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MT + DN (Experimental): 4 treatment sessions of 20 minutes manual therapy will be given over 4 weeks (1session/week). The techniques will be tailored to the patients needs, and will exclude 'High Velocity Low Amplitude' manipulations.
  In addition, a maximum of 4 muscles will be treated by means of dry needling in at least 3 sessions, based on the pain pattern of the patient.
  Interventions: Other: Dry Needling; Other: Manual therapy
- MT alone (Active Comparator): 4 treatment sessions of 20 minutes manual therapy will be given over 4 weeks (1session/week). The techniques will be tailored to the patients needs, and will exclude 'High Velocity Low Amplitude' manipulations.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Dry Needling — Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increase in blood flow,recovery of the muscle metabolism and thus a reduction of pain and stiffness.
  Arms: MT + DN
Other: Manual therapy — Manual therapy comprises stretching of muscles, mobilizations, traction and translation of vertebrae, Sustained Natural Apophyseal Glides (SNAG), dynamic soft tissue mobilization, Muscle Energy Techniques (MET) and home-exercises.

SUMMARY:
This project comprises two studies; a cross-sectional study and a randomized controlled trial.

1. The goal of the cross-sectional study is to compare multiple outcome parameters in different headache types: tension type (TTH), cervicogenic (CGH) and myofascial headache (MFH) as drafted by the International Classification of Headache Disorders (ICHD). Not only will these types be compared against each other, they will also be compared to healthy controls (HC).

   The main research questions are:
   * Are the criteria drafted by the International Classification of Headache Disorders (ICHD) discriminative for MFH?
   * Are there differences between the headache types (and healthy controls) in pain & disability scores, range of motion (ROM), muscle strength, muscle elasticity and hyperalgesia (=pain pressure threshold, PPT)?

   Participants will :
   * Fill out questionnaires about their pain and disability;
   * Be clinically investigated by a physiotherapist (anamnesis, inspection, examination of movement and structures of the neck and head);
   * Undergo a testing battery including neck ROM, neck muscle strength & elasticity and PPT measurement of the C2 processus spinosus, the bilateral upper trapezius muscle and the tibialis anterior muscle of the dominant leg.
2. The goal of this randomized controlled study is to investigate the additional effect of dry needling in the treatment of MFH patients, as compared to a treatment consisting of manual techniques only. The main question it aims to answer is:

   * Does manual therapy combined with dry needling provide an additional effect on pain, disability and functional outcomes in MFH patients, as compared to manual therapy alone?

After the baseline test (see part 1), participants with MFH will be randomly divided to receive 4 sessions over 4 weeks of MT or MT + DN. Hereafter, the baseline test is repeated at 1 week and 3 months post-treatment.

DETAILED DESCRIPTION:
Although tension-type headache (TTH) and cervicogenic headache (CGH) are classified as two distinct headache types according to the International Classification of Headache Disorders (ICHD), there are many cases in which overlap between these two types exists, and for whom clinical diagnosis can be challenging. Peripheral activation or sensitization of myofascial nociceptors is suggested as a potential mechanism in both categories, and as a consequence the ICHD (3rd edition - 2018) has recently drafted an alternative diagnosis: headache attributed to cervical myofascial pain (MFH). However, clear clinical criteria for this diagnosis are currently lacking.

By subjecting CGH, TT, MFH and HC (34 participants of each) to the ICHD criteria and a clinical investigation, we will look at similarities and differences and the ability of the criteria to differentiate the headache types.

Among the several proposed approaches for the treatment of myofascial pain, dry needling (DN) has received particular attention in the last decades. DN is defined as a skilled intervention using a thin needle which is inserted into a painful point in the muscle, also referred to as a trigger point. Although previous studies have indicated that DN may be an effective intervention in the treatment of TTH and CGH, little is known about its (additional) effect on MFH.

Therefore, 50 MFH patients will be recruited. Participants are included based on online questionnaires, a clinical examination of the neck and the ICHD criteria. All participants will receive information and have to sign an informed consent form. Participants will be subjected to baseline assessment, which involves measurements of pain scores (NPRS), hyperalgesia (PPT by algometry), ROM (EasyAngle device) and neck muscle strength measurement (EasyForce device) and neck muscle elasticity measurement using Shear Wave Elastography (SWE). Then, participants will be randomly allocated to either a manual therapy group or a manual therapy + dry needling group. 4 sessions of therapy will be given over 4 weeks time.

1 week and 3 months after the treatment sessions, the baseline measurements will be repeated. After 6 and 12 months, patients will complete questionnaires from home which will give information about pain & disability scores.

.

ELIGIBILITY:
Inclusion Criteria:

* < 15 headache days per month
* > 5 episodes of the headache that gives hindrance
* Mean NPRS score for headache episodes >2/10
* No history of whiplash
* No serious structural pathology
* No previous surgeries in the head/neck/shoulder region

To be included in the RCT-part of the study:

- Fitting the ICHD criteria for MFH

Exclusion Criteria:

* Diagnosis of migraine by a neurologist or as confirmed via the Headache Screening Questionnaire (HSQ) with the maximum score of 8/8.
* Chronic headache (>15 headache days/month)
* Newly onset headache (<5 previous episodes of new headache type)
* Whiplash or whiplash associated disorders
* Serious structural pathology (confirmed by medical imaging)
* Pain on both sides of the body, above and under the waist, (with a total score of 7 or more out of 10) (=Widespread pain)
* Cardiovascular/metabolic/systemic/neurological diseases
* Fibromyalgia, Chronic Fatigue Syndrome
* History of surgery in the head/neck or shoulder region
* Probable or definite neuropathic pain (according to the classification of Finnerup et al.)
* Traumatic onset of the complaints
* Pregnancy/given birth/breastfeeding in the preceding year
* Psychiatric illnesses or depression diagnosed by a psychiatrist and currently treated by a psychiatrist and/or medication.
* BMI >30

For all of RCT-patients, the following criteria will also lead to exclusion due to the dry needling intervention:

* Usage of heavy blood thinners or anti-coagulants (e.g. Marcoumar, Marevan, Sintrom)
* High risk of infection because of comorbidities (e.g. HIV, diabetes) or skin conditions in the neck region (e.g. psoriasis)
* Epilepsy
* Allergies for latex, nickel
* Needle phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Headache Disability Inventory (HDI) | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  The HDI is a 25-item questionnaire of which the questions focus on two categories. There are 13 questions related to the emotional effects and 12 questions on the functional effects of headache complaints. There are 3 answer options: yes (4 points), sometimes (2 points), no (0 points). The sum (maximum 100) gives an impression about the self-perceived limitations as a result of headache. The higher the score, the greater the hindrance caused by headache.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  Changes in neck disability scores will be assessed by the Neck Disability Index. The Neck Disability Index consists of 10 questions, each with 6 answer options with concomitant scores ranging from 0 to 5, which makes the total score of the NDI on 50. A score between 5 and 14 represents a mild disability, whereas a score between 15 and 24 is interpreted as a moderate disability. NDI scores of 25 or higher reflect a severe disability.
Numeric Pain Rating Scale (NPRS) | Baseline; right before each treatment session; 1 week, 3 months, 6 months, 12 months post-treatment
  Patient's neck pain and headache will be measured using an 11-point NRS, with a minimum value of zero ("no pain") and a maximum score of 10 ("the worst pain possible")
Range of Motion (ROM) | Baseline; 1 week and 3 months post-treatment
  Using the EasyAngle device (Meloq Instruments), patients' neck ROM will be measured from a sitting position. Each movement (flexion, extension, bilateral lateral flexion and bilateral rotation) will be performed thrice. This will be done by the same researcher at every test moment.
Muscle strength (Fm) | Baseline; 1 week and 3 months post-treatment
  Using the EasyForce device (Meloq Instruments), patients' neck muscle strength will be measured from a sitting position for lateral flexion (bilaterally) or from a supine or prone lying position for neck flexion and extension respectively. Three trials of 5 seconds of maximal force will be executed with 30 seconds rest between them. This will be guided by the same researcher at every test moment.
Pressure Pain Threshold (PPT) | Baseline; 1 week and 3 months post-treatment
  To measure local and distal hyperalgesia, a digital handheld pressure algometer (FDX; Wagner Instruments) will be used on the C2 processus spinosus, both upper trapezius muscles and the M. Tibialis Anterior of the dominant leg.
  To measure the PPT, the researcher will apply the digital algometer to each of the indicated points with a round rubber end of 1 cm² and an increasing pressure of circa 1 kgf/s. As soon as the sensation of the subject shifts from a comfortable pressure to an altered, unpleasant feeling, the participant reports this and the test will be finished.
  Each point will be measured three times with a 30-second interval in between and all measurements will be performed by one researcher in the same standardised position for each point.
Muscle Elasticity | Baseline; 1 week and 3 months post-treatment
  For measuring the patients' muscle elasticity, Shear Wave Elastography (SuperSonic Imagine S.A., Aix-en-Provence, France) will be used.From supine lying, M. Sternocleidomastoideus and M. Masseter will be measured, whereas M. Trapezius pars descendens & ascendens, M. Splenius Capitis & Cervicis and M. Semispinalis Capitis & Cervicis will be measured from prone lying. Measurements will be made after 10 minutes of lying down and relaxing. Of each muscle, 3 recordings of 15 seconds will be taken bilaterally. This will always be performed by the same researcher.
Global Perceived Effect (GPE) | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  Changes in Global Perceived Effect scores as assessed by the Global Perceived Effect Scale. This scale consists of 7 scores (ranging from 1 (a lot better) to 7 (a lot worse)).
Headache Impact Test (HIT-6) | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  Headache related disability will be questioned using the Headache Impact Test (HIT-6) questionnaire. The total score can range from 36 to 78, with a higher score indicating the headache has more impact on daily life.
Central Sensitization Index (CSI). | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  The Central Sensitization Index (CSI) score ranges from 0 to 100, allowing to make the following classifications of sensitization:
  0-29 Subclinical 30-39 Mild 40-49 Moderate 50-59 Severe 60-100 Extreme
Pain Catastrophizing Scale (PCS) | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  The Pain Catastrophizing Scale (PCS) has 13 items, each belonging to one of three of the following subscales:
  * Rumination (item 8,9,10,11)
  * Magnification (item 6,7,13)
  * Helplessness (item 1,2,3,4,5,12) The total score of the questionnaire ranges from 0 to 52. The higher the score, the more pain catastrophizing the patient shows.
Pain Coping Inventory(PCI). | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  The Pain Coping Inventory (PCI) records which coping strategy is preferred by the patient. The inventory contains 6 scales which can be divided in active coping strategies (Pain Transformation, Distraction, Reducing Demands) or passive coping strategies (Retreating, Worrying, Resting).
  The higher the score per domain, the more the patients uses that type of coping.
Tampa Scale of Kinesiophobia (TSK). | Baseline; 1 week, 3 months, 6 months, 12 months post-treatment
  The Tampa Scale of Kinesiophobia (TSK) contains 17 items and the total score can range from 17 to 68.
  A score of more than 37 points towards kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Universitair ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The website will depend on the journal in which the sponsor will publish